CLINICAL TRIAL: NCT06573268
Title: One-year Clinical Experiences of Single-port and Multi-port Robotic Thyroid Surgery in Single Institution
Brief Title: Da-vinci sp Versus xi Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Jin Wook Yi, Associate Professor, Inha University Hospital
Other Study IDs: 2024-08-015
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Cancer; Thyroid Nodule
Keywords: thyroid; robotic surgical procedures; minimally invasive surgical procedures
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Nodule; Thyroid Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SPRA: patients who received da-Vinci SP robot thyroid surgery by SPRA method (Single Port Robotic Areolar)
  Interventions: Device: robot surgery device
- BABA: patients who received da-Vinci SP robot thyroid surgery by BABA method (Bilateral Axillary Breast Approach)
  Interventions: Device: robot surgery device

INTERVENTIONS:
Device: robot surgery device — SPRA used da-Vinci SP system (SPRA) BABA used da-Vinci Xi system (BABA)

SUMMARY:
One year comparative analysis between SPRA* versus BABA** thyroid surgery. * SPRA: da-Vinci SP Robotic Areolar approach thyroid surgery

** BABA: da-Vinci Xi robotic Bilateral. Axillary Breast Approach thyroid surgery

DETAILED DESCRIPTION:
Study design: retrospective data analysis Study period: December 2022 to December 2023 Candidate: Patients who received robot thyroid surgery during study period Numbers of candidates: total of 270 patients Group : SPRA (n=111) versus BABA (n=159) Statistic analysis: t-test for continuous variable, fisher's exact test for categorical variable

ELIGIBILITY:
Inclusion Criteria:

* Patients who received robot thyroid surgery in our institution
* Retrospective review

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received robot thyroid surgery in our institution during study period
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Total operation time (minutes) | on the surgery day (1 day)
  Time for spending total surgery

SECONDARY OUTCOMES:
Hospital stay days after surgery | after the surgery day (up to 2 weeks)
  Hospital admission days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Choi YS, Choi JH, Jeon MS, Yu MJ, Lee HM, Shin AY, Yi JW. First Experience of Single-Port Robotic Areolar Approach Thyroidectomy. Clin Exp Otorhinolaryngol. 2023 Aug;16(3):275-281. doi: 10.21053/ceo.2023.00682. Epub 2023 Jul 5. PMID 37475141
- [Result] Choi YS, Shin WY, Yi JW. Single Surgeon Experience with 500 Cases of the Robotic Bilateral Axillary Breast Approach (BABA) for Thyroid Surgery Using the Da-Vinci Xi System. J Clin Med. 2021 Sep 7;10(18):4048. doi: 10.3390/jcm10184048. PMID 34575159